CLINICAL TRIAL: NCT01651650
Title: An Open Label Placebo Study to Assess the Inhalation Profile in Asthmatic Patients Using the Nexthaler® Dry Powder Inhaler (DPI) Device
Acronym: NEXThalerPIF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCD-1113-PR-0074; 2012-000039-22 (EudraCT Number)
Record Dates: First submitted 2012-07-05; First posted 2012-07-27 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2017-03

CONDITIONS: Asthma
Keywords: Asthma; PIF
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inhalation of Placebo Dry Powder (Other): Each patient will perform at least two inhalations using the Chiesi NEXThaler DPI device containing placebo dry powder. There is no comparator and all patients will receive the same study treatment.
  Interventions: Device: Inhalation through Chiesi NEXThaler DPI

INTERVENTIONS:
Device: Inhalation through Chiesi NEXThaler DPI — Inhalatory manoeuvre through Chiesi NEXThaler DPI repeated at least twice in order to have two evaluable data set

SUMMARY:
Phase IIa, single-centre, open-label, single-arm study, to evaluate the inspiration profile through the NEXThaler® device in adult asthmatic patients with varying degrees of disease control.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the inspiratory flow profile through the NEXThaler® device in adult asthmatics with varying degrees of disease control.

The study plan foresees one visit at clinic. At Visit 1, after the signature of the informed consent form, the inclusion/exclusion criteria will be checked and the lung function parameters will be evaluated. If the subjects meet the inclusion/exclusion criteria, they will be instructed to use the NEXThaler®. The patients will subsequently inhale through the device and the inspiration profile will be measured.

A total of 40 asthmatic adults (≥18 years), 20 with controlled stable disease and 20 with partly controlled or uncontrolled disease according to GINA guidelines (2011), will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of controlled, partly controlled or uncontrolled asthma according to GINA guidelines (2011)
* A cooperative attitude and ability to use DPIs and to be trained in the proper use of the NEXThaler® as confirmed by the activation of the training device BAM

Exclusion Criteria:

* Significant seasonal variation in asthma or asthma occurring only during episodic exposure to an allergen or a chemical sensitizer
* History of near fatal asthma (e.g. brittle asthma, hospitalisation for asthma exacerbation in Intensive Care Unit)
* Diagnosis of restrictive lung disease
* Significant unstable medical history of and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any laboratory abnormality indicative of a significant underlying condition, that may interfere with patient's safety, compliance, or study evaluations, according to the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of inhalatory profile for 40 patients | One visit per patient (visit 1)
  The study duration per patient is only one visit. At visit 1 the patient after having signed off the ICF and after having assessed the Eligibility Criteria should perform two evaluable inhalatory manoeuvres. Each manoeuvre lasts few seconds. After having completed the manoeuvres and have the same assessed as good by the Investigator, the study is completed. All the procedures are expected to be performed within a couple of hours for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo A. Chetta, MD, Principal Investigator — Clinica Pneumologica, AOU di Parma
Locations (1):
- Clinica Pneumologica, AOU di Parma, Parma, Italy

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2012-000039-22